CLINICAL TRIAL: NCT04428021
Title: Effectiveness of Adding Standard Plasma or COVID-19 Convalescent Plasma to Standard Treatment, Versus Standard Treatment Alone, in Patients With Recent Onset of COVID-19 Respiratory Failure. A Randomized, Three-arms, Phase 2 Trial
Brief Title: Standard or Convalescent Plasma in Patients With Recent Onset of COVID-19 Respiratory Failure
Acronym: PLACO-COVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Paola Maria Manzini, Principal Investigator, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CS3/33
Record Dates: First submitted 2020-06-07; First posted 2020-06-11 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Three arms randomized trial, partially blinded
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Only the two experimental arms are masked. COVID-19 convalescent plasma (CP) and standard plasma (SP) will be masked and delivered to the wards in identical bags; a tag printed as "PLASMA TRIAL" will cover the actual name of the product
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard therapy protocol (STP) (Active Comparator): STP is defined as the best evidence based therapy approved for treatment of COVID-19 patients by Regional Health System emergency committee. STP could be updated during the trial.
  Interventions: Drug: Standard Therapy Protocol (STP)
- STP + Standard Plasma (SP) (Experimental): STP + 3 units on day 1-3-5 of Standard Plasma collected in pre-COVID era (January-September 2019)
  Interventions: Drug: Standard Therapy Protocol (STP); Other: STP + Standard Plasma (SP)
- STP + COVID-19 Convalescent Plasma (CP) (Experimental): STP + 3 units on day 1-3-5 of COVID-19 Convalescent Plasma containing neutralizing SARS-Cov-2 antibodies
  Interventions: Drug: Standard Therapy Protocol (STP); Other: STP + COVID-19 Convalescent Plasma (CP)

INTERVENTIONS:
Drug: Standard Therapy Protocol (STP) — Standard Therapy Protocol according to the best evidence treatment recommended by the Regional Health System emergency committee
Other: STP + Standard Plasma (SP) — Transfusion of three Standard Plasma Units (SP) on day 1,3,5 in addition to STP
  Arms: STP + Standard Plasma (SP)
Other: STP + COVID-19 Convalescent Plasma (CP) — Transfusion of three SARS-Cov-2 neutralizing antibodies positive Plasma Units (CP) on day 1,3,5 in addition to STP
  Arms: STP + COVID-19 Convalescent Plasma (CP)

SUMMARY:
To date no specific treatment has been proven to be effective for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-Cov-2) infection. It is possible that convalescent plasma that contains antibodies to SARS-Cov-2 might be effective against the progression of infection. Promising results have been shown by preliminary data from China cases. The investigators planned to compare effectiveness of adding COVID-19 convalescent plasma to standard therapy protocol (STP) versus adding plasma donated in pre-COVID era versus STP alone in patient with COVID-19 within 5 days from the onset of respiratory distress. STP at enrolment is the best evidence based therapy approved for treatment of COVID patients by regional Health system emergency committee.

DETAILED DESCRIPTION:
500-700 ml of Plasma will be collected by apheresis from COVID recovered donors showing the presence of neutralizing antibodies to SARS-Cov-2 (anti-SARS-Cov-2). All plasma will be screened for transmissible diseases according to italian law (Hepatitis B Virus,Hepatitis C Virus, Human Immunodeficiency Virus 1-2, Syphilis) plus adjunctive screening for Hepatitis A Virus and Hepatitis E Virus-RNA and Parvovirus B19-DNA as requested from Italian National Blood Authority. Apheresis will be divided in two/three units (170-300 ml each), virus inactivated with Riboflavin and ultraviolet light illumination technology and immediately frozen and stored separately from other plasma bags.

Enrolled patients will be stratified according to severity of respiratory failure and randomized in three arms: 1) Standard Therapy Protocol (STP), 2) Standard Therapy Protocol + 170-350 ml standard Plasma (SP) on day 1-3-5 after randomization, 3) Standard Therapy Protocol + 170-350 ml COVID-19 Convalescent Plasma on day 1-3-5 after randomization.

The three therapeutic units of COVID-19 Convalescent plasma will be chosen in order to minimize variations among patients in the total amount of infused SARS-Cov-2 antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed SARS-Cov-2 diagnosis by RT-PCR on nasopharyngeal swab or on bronchoalveolar lavage
* Respiratory failure onset or progression within 5 days
* Signed Informed Consent

Exclusion Criteria:

* Pregnancy
* Previous severe reactions to plasma transfusion
* Unavailability of blood group compatible COVID-19 convalescent plasma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
30-days survival | 30 days after randomization
  Proportion of patients alive 30 days after randomization

SECONDARY OUTCOMES:
Ventilator free survival | 30 days after randomization
  Cumulative incidence of mechanical ventilation or death
6-months survival | 6 months after randomization
  Probability of being alive at 6 months after randomization
Incidence of complications | Within 12 months
  Proportion of patients developing any serious medical or procedure related complications
Days in intensive care units (ICU) | From date of randomization until the date of discharge or date of death from any cause, whichever came first, assessed up to 12 months
  Proportion of days spent in ICU on the total length of hospital stay
Positivity for Immunoglobulin G to SARS-Cov-2 | On day 0, 2, 4, 6,10,14, 21, 28 after randomization and at date of discharge or death from any cause, whichever came first, assessed up to 12 months
  Proportion of patients showing seroconversion to Immunoglobulin G (IgG) anti-SARS-Cov-2
Clearance of viral load | On day 0, 2, 4, 6,10,14, 21, 28 after randomization and at date of discharge or death from any cause, whichever came first, assessed up to 12 months
  Proportion of patients showing viral clearance by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) on plasma and respiratory tract samples
Sequential Organ Failure Assessment (SOFA) score | On day 0, 2, 4, 6, 10, 14, 28 after randomization and at date of discharge or death from any cause, whichever came first, assessed up to 12 months
  Variations in SOFA Score (range 0-24; higher score mean a worse outcome)
Any variation from Standard Therapy Protocol | From date of randomization until the date of discharge or date of death from any cause, whichever came first, assessed daily up to 2 months
  Proportion of patients needing introduction of new drug or discontinuation of drug from standard therapy protocol

CONTACTS AND LOCATIONS:
Overall Officials: Paola Maria Manzini, MD, Principal Investigator — AO Città della salute e della scienza di Torino
Locations (1):
- AO Città della salute e della scienza di Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: Yes
All Individual Participant Data requests should be submitted to the corresponding author for consideration. Access to deidentified participant data may be granted following review, after the publication of major results
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available after 12 months from study ending and for the following 5 years
Access Criteria: Data requests should be submitted to the corresponding author for consideration.

REFERENCES:
- [Derived] Manzini PM, Ciccone G, De Rosa FG, Cavallo R, Ghisetti V, D'Antico S, Galassi C, Saccona F, Castiglione A, Birocco N, Francisci T, Hu H, Pecoraro C, Danielle F, Labanca L, Bordiga AM, Lorenzi M, Camisasca G, Giachino O, Pagliarino M, Ottone P, Scuvera ITD, Guaschino R, Freilone R, Berti P, Pittaluga F, Avolio M, Costa C, Raso S, Nucci A, Milan M, Baffa A, Russo A, Tornello A, Maddalena L, Delios G, Marletto FP, De Micheli AG, Mattei A, Baldassano S, Canta F, Russo ML, Bergamo D, Vitale F, Liccardi MM, Chinaglia A, Calcagno A, Converso M, Aldieri C, Libanore V, Blangetti I, Benedetti V, Mitola B, Scozzari G; PLACO COVID Study Group. Convalescent or standard plasma versus standard of care in the treatment of COVID-19 patients with respiratory impairment: short and long-term effects. A three-arm randomized controlled clinical trial. BMC Infect Dis. 2022 Nov 22;22(1):879. doi: 10.1186/s12879-022-07716-5. PMID 36418984